CLINICAL TRIAL: NCT06008873
Title: Association Between Preoperative Insomnia and Postoperative Quality of Recovery in Non-elderly Patients Undergoing Non-emergency Cancer Resection Surgery: A Prospective Observational Study
Brief Title: Association Between Preoperative Insomnia and Postoperative Quality of Recovery : A Prospective Observational Study
Acronym: PIPQoR
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2023ZSLYEC-260
Record Dates: First submitted 2023-08-13; First posted 2023-08-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disorder
Keywords: Insomnia; Perioperative Medicine; cancer; surgery; Quality of Recovery
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- One group only: No intervention.

SUMMARY:
Although patients with cancers are prone to insomnia, especially waiting for surgery during hospitalization, and insomnia promotes acute respiratory infections (ARI) and is not conducive to the postoperative quality of recovery (QoR), evidence that preoperative insomnia delays postoperative recovery is still lacking. In this prospective observational study, we enroll 175 non-elderly subjects with abdominal cancer who will undergo non-emergency cancer resection surgery. Insomnia Severity Index scale (ISI) is used to assess the insomnia severity during hospitalization while awaiting surgery. The Quality of Recovery-15 (QoR-15) is used to evaluate the overall recovery after surgery. Meanwhile, wrist watch and sleep diary are used to record sleep. The aim of the study is to investigate the association between preoperative insomnia and postoperative QoR, the association between preoperative insomnia and postoperative ARI,and to describe preoperative sleep traits.

DETAILED DESCRIPTION:
In the single-center, prospective observational study, ISI is used to investigate the perceptive sleep during hospitalization waiting for surgery,and QoR-15 is used to investigate the overall quality of functional recovery at postoperative 1, 3, 7, 14, and 30 days (POD1/3/7/14/30). At the same time, both of ARI within POD30 and neutrophil to lymphocyte ratio(NLR) in peripheral blood perioperation are recorded. The study is divided into four phases: (1) Screening: on the first day of admission, the subjects are screened according to the inclusion and exclusion criteria, and the basic data are collected, including ISI, QoR-15 and depression/anxiety questionnaires, et al. (2) Enrollment (sleep survey during hospitalization waiting for surgery) : ISI is performed in the day of surgery to perceive the severity of insomnia during the whole period of hospitalization waiting for surgery, and objective and subjective sleep are investigated by wrist watch and sleep diary. (3) Surgical and anesthesia period: the key medical data related to surgery, anesthesia and nursing occurred during the operation are recorded. (4) Follow-up: QoR-15 is investigated POD1/3/7/14/30. Meanwhile, both of ARI and NLR are investigated.

The planned enrollment is 175 subjects. No randomized or any protocol-driven treatment is administered to the subjects during the study. The effect size f2 of the independent variable (ISI scores of hospitalization waiting for surgery) on the dependent variable (QoR-15 on POD1) is expected to be 0.1. The number of covariates is predicted to be 46, α is set as two-sided 0.05, and the power is 0.9. The sample size calculated by PASS software is 157 cases. Considering 10% dropout, a sample size of 175 will be required. Data will be presented as mean±standard deviation, median and number (%). Logistic multivariate, or multivariable models will be both performed by statisticians.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntarily execute informed consent;
* 2.Effective linguistic communication and collaboration;
* 3.No history of mental disorders;
* 4.Age of 18-64 years old, male or female;
* 5.BMI 18-30kg/m2;
* 6.American Society of anesthesiology (ASA) grade 1-2, New York Heart Association(NYHA) grade Ⅰ or Ⅱ;
* 7.Initial diagnosis of abdominal cancers and the diagnosis has been disclosed to subjects;
* 8.Non-emergency cancer resection surgery is planned;
* 9.The planned anesthesia is general anesthesia with endotracheal intubation.

Exclusion Criteria:

* 1.Obstructive apnea syndrome, narcolepsy, restless leg/periodic limb movement disorder, sleepwalking disorder, nightmare disorder;
* 2.Not suitable to participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Referred to the Eligibility Criteria for details.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Total scores of the questionnaire of Insomnia Severity Scale (ISI) on the day before surgery or the day of surgery | on the day before surgery or the day of surgery
  ISI is used to assess insomnia during the time when waiting for surgery in hospital from the day of admission to the day of surgery.
  ISI is used to assess how satisfied with sleep patterns and psychological distress or impairments in daytime functioning associated with sleep difficulties.
  ISI is filled in by subjects on the day before surgery or the day of surgery. ISI contents 7 items, which item is measured by an 0-4 point rating scale (0="very satisfaction"; 4="very dissatisfaction").
  ISI total scores range from 0 to 28, with higher scores indicating higher severity of insomnia.
Total scores of the questionnaire of 15-item Quality of Recovery scale (QoR-15）on postoperative day 1 | on postoperative day 1
  QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically.
  QoR-15 is filled on postoperative day 1. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0= "none of the time" to 10="all of the time"; for negative items the scoring was reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).

SECONDARY OUTCOMES:
Sleep-onset latency(min)(resulting from CSD): Distribution frequency of different degrees of sleep latency during the time when waiting for surgery in hospital from the day of admission to the day of surgery | Everyday when waiting for surgery in hospital from the day of admission to the day of surgery
  A Consensus Sleep Diary (CSD) is used to asses subjective sleep quantity everyday when waiting for surgery in hospital from the day of admission to the day of surgery.
  The CSD items assess sleep-onset latency (time taken to fall asleep), the number of awakenings, and the total duration of sleep. Subjects also allow to record factors that could influence sleep, including use of sleep medication.
Numbers of awakenings(resulting from CSD): Distribution of Numbers of awakenings during the time when waiting for surgery in hospital from the day of admission to the day of surgery | Everyday when waiting for surgery in hospital from the day of admission to the day of surgery
  A Consensus Sleep Diary (CSD) is used to asses subjective sleep quantity everyday waiting for surgery in hospital from the day of admission to the day of surgery.
  The CSD items assess sleep-onset latency (time taken to fall asleep), the number of awakenings, and the total duration of sleep. Subjects also allow to record factors that could influence sleep, including use of sleep medication.
Total duration of sleep in night(min)(resulting from CSD): Distribution of total duration of sleep in night during the time when waiting for surgery in hospital from the day of admission to the day of surgery | Everyday when waiting for surgery in hospital from the day of admission to the day of surgery
  A Consensus Sleep Diary (CSD) is used to asses subjective sleep quantity everyday waiting for surgery in hospital from the day of admission to the day of surgery.
  The CSD items assess sleep-onset latency (time taken to fall asleep), the number of awakenings, and the total duration of sleep. Subjects also allow to record factors that could influence sleep, including use of sleep medication.
Sleep influencing factors(resulting from CSD): Distribution of factors that could influence sleep in night when waiting for surgery in hospital from the day of admission to the day of surgery | Everyday when waiting for surgery in hospital from the day of admission to the day of surgery
  A Consensus Sleep Diary (CSD) is used to asses subjective sleep quantity everyday waiting for surgery in hospital from the day of admission to the day of surgery.
  The CSD items assess sleep-onset latency (time taken to fall asleep), the number of awakenings, and the total duration of sleep. Subjects also allow to record factors that could influence sleep, including use of sleep medication.
Total scores of the questionnaire of 15-item Quality of Recovery scale (QoR-15）on postoperative day 3 | on postoperative day 3
  QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically.
  QoR-15 is filled on postoperative day 1. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0= "none of the time" to 10="all of the time"; for negative items the scoring was reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Total scores of the questionnaire of 15-item Quality of Recovery scale (QoR-15）on postoperative day 7 | on postoperative day 7
  QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically.
  QoR-15 is filled on postoperative day 1. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0= "none of the time" to 10="all of the time"; for negative items the scoring was reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Total scores of the questionnaire of 15-item Quality of Recovery scale (QoR-15）on postoperative day 14 | on postoperative day 14
  QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically.
  QoR-15 is filled on postoperative day 1. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0= "none of the time" to 10="all of the time"; for negative items the scoring was reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Total scores of the questionnaire of 15-item Quality of Recovery scale (QoR-15）on postoperative day 30 | on postoperative day 30
  QoR-15 is a patient-reported measure, and is used to assess global recovery quality after surgery physiologically and psychologically.
  QoR-15 is filled on postoperative day 1. QoR-15 contents 15 items, which item is constructed by an 11-point numerical rating scale (for positive items, 0="none of the time" to 10="all of the time"; for negative items the scoring was reversed). The total scores are ranging from 0(extremely poor QoR) to 150 (excellent QoR).
Incidence rate of Acute Respiratory Tract Infection (ARTI) within postoperative day 30 | within postoperative day 30
  Acute Respiratory Tract Infection (ARTI): including acute upper respiratory infection and acute lower respiratory infection, according to patients self-reporting.
Peripheral blood neutrophil/lymphocyte ratio on postoperative day 1 | on postoperative day 1
  Peripheral blood neutrophil/lymphocyte ratio on postoperative day 1 resulting from blood routine examination
Peripheral blood neutrophil/lymphocyte ratio on postoperative day 3 | on postoperative day 3
  Peripheral blood neutrophil/lymphocyte ratio on postoperative day 3 from blood routine examination
Peripheral blood neutrophil/lymphocyte ratio on postoperative day 7 | on postoperative day 7
  Peripheral blood neutrophil/lymphocyte ratio on postoperative day 7 from blood routine examination

CONTACTS AND LOCATIONS:
Overall Officials: Jin sanqing, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No